CLINICAL TRIAL: NCT01313351
Title: A Clinical Evaluation of the RPS InflammaDry Detector's Sensitivity and Specificity Compared to the Clinical Diagnosis for Confirming Dry Eyes.
Brief Title: RPS InflammaDry Detector™ to Determine MMP-9 Levels in Tears
Status: Completed | Type: Observational
Sponsor: Rapid Pathogen Screening (Industry)
Responsible Party: Sponsor
Organization: Lumos Diagnostics (Industry)
Other Study IDs: 100310
Record Dates: First submitted 2011-03-03; First posted 2011-03-11 (Estimated); Results first posted 2022-03-16 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-11

CONDITIONS: Dry Eye
Keywords: Dry eyes; Dysfunctional tear syndrome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Device testing: Tears were collected from subjects to apply to the RPS InflammaDry detector and were clinically evaluated.
  Interventions: Device: RPS InflammaDry Detector™

INTERVENTIONS:
Device: RPS InflammaDry Detector™ — A noninvasive immunoassay for detecting MMP-9 levels in tears

SUMMARY:
The RPS InflammaDry Detector™ is intended to detect elevated MMP-9 in human tears to aid in the diagnosis of patients with signs or symptoms of dry eye disease, in conjunction with other methods of clinical evaluation.

DETAILED DESCRIPTION:
The purpose of this clinical trial was to determine the sensitivity and specificity of InflammaDry compared with the clinical assessment of dry eyes.

Patients were screened using clinical history and signs.

Clinical history was performed using the Ocular Surface Disease Index (OSDI) and evaluated for clinical signs:

* positive vital staining of the ocular surface,
* decreased tear breakup time (TBUT),
* reduced corneal sensitivity, and
* decreased functional visual acuity Last, an independent health care professional masked to the clinical evaluation was asked to analyze each InflammaDry test result, independently confirming each result.

ELIGIBILITY:
INCLUSION CRITERIA

Patients older than 18 years of age, who meet the following criteria related to the clinical history and signs will be enrolled:

Group 1: Clinical Dry Eyes

Clinical History Criteria

An Ocular Surface Disease Index (OSDI) of greater than or equal to 13 - [Appendix #2]

Clinical Signs Criteria - All of the following must be present

1. Schirmer's Tear Test (with anesthesia) < 10 mm over 5 minutes
2. Tear Film Break Up Time (TBUT) < 10 seconds
3. Total Corneal Staining ≥ 1 [Appendix #1]

   * At least 1/2 of all patients enrolled will have a Schirmer's Tear Test < 5 mm or demonstrate corneal staining ≥ 2 [Appendix #1]

Group 2: Clinical Normal Non-Dry Eyes

Clinical History Criteria

An Ocular Surface Disease Index (OSDI) of < 7 - [Appendix #2]

Clinical Signs Criteria - All 3 of the following must be present

1. Schirmer's Tear Test (with anesthesia) ≥ 10 mm over 5 minutes
2. Tear Film Break Up Time (TBUT) ≥ 10 seconds
3. Total Corneal Staining = 0 [Appendix #1]

EXCLUSION CRITERIA

* Patients with allergy to corn starch, talcum powder, or dacron
* Patients with prior eye injury, trauma, or ocular surgery within the previous 3 months
* Patients with non-dry eye ocular inflammation, uveitis, history of herpetic keratitis or zoster keratitis
* Patients with history of a recent ocular infection within the prior 1 month
* Use of oral doxycycline or topical macrolides (AzaSite) within 1 month
* Patients currently receiving, or received in the last 2 weeks of the study , certain medications including topical or systemic corticosteroids, topical or systemic Nonsteroidal (NSAIDs) therapy, topical cyclosporine, or other immunosuppressive therapy
* Patients who are pregnant or lactating
* Before initialization of the study, patients must not have used any topical medications, including artificial tears during the previous 2 hours
* The use of Rigid-Gas permeable contact lenses or the use of soft-contact lenses within 1 month of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Only patients who met the inclusion criteria were included in the study.
Sampling Method: Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2010-11; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sambursky, MD, Study Director — Rapid Pathogen Screening, Inc.
Locations (8):
- United States (8):
  - Manatee Sarasota Eye Clinic, Bradenton, Florida
  - Center for Excellence in Eye Care, Miami, Florida
  - St. John's Clinics, Springfield, Missouri
  - Ophthalmic Consultants of Long Island, Lynbrook, New York
  - Physician Eyecare of NY, New York, New York
  - Weill-Cornell Medical College, New York, New York
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - William F. Davitt, III, MD, El Paso, Texas

REFERENCES:
- [Derived] Sambursky R, Davitt WF 3rd, Latkany R, Tauber S, Starr C, Friedberg M, Dirks MS, McDonald M. Sensitivity and specificity of a point-of-care matrix metalloproteinase 9 immunoassay for diagnosing inflammation related to dry eye. JAMA Ophthalmol. 2013 Jan;131(1):24-8. doi: 10.1001/jamaophthalmol.2013.561. PMID 23307206

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Device Testing
Started | 206
Completed | 206
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- InflammaDry Test: Tears were collected from subjects to apply to the RPS InflammaDry detector and were clinically evaluated.
  RPS InflammaDry Detector™: A noninvasive immunoassay for detecting MMP-9 levels in tears
Arm/Group | InflammaDry Test
Number analyzed (Participants) | 206
Age, Continuous [Mean (Full Range); unit: years] | 53 [18 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152
  Male | 54
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 136
  Race: Black | 11
  Race: Hispanic | 49
  Race: Asian | 9
  Race: Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 206

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity and Specificity of InflammaDry Detector Compared to Clinical Assessment at Confirming a Diagnosis of Dry Eyes.
Description: Patients were assessed for signs and Symptoms of Dry Eye using OSDI (Ocular Surface Disease Index), TBUT (Fluorescein Tear Break-up Time), Corneal fluorescein staining and Schirmer Tear Test and compared to the results of the tested device.
  Sensitivity is the percentage of true positive cases correctly identified by the test, compared to clinical assessment.
  Specificity is the percentage of true negative cases correctly identified by the test, compared to clinical assessment.
Time Frame: 15 minutes
Measure: Number (95% Confidence Interval); unit: percentage of cases
Groups:
- InflammaDry Sensitivity: Percentage of True Positives when compared to Clinical Assessment
- InflammaDry Specificity: Percentage of True Negatives when compared to Clinical Assessment
Arm/Group | InflammaDry Sensitivity | InflammaDry Specificity
Number analyzed (Participants) | 143 | 63
percentage of cases | 85 [77.6 to 90.5] | 94 [84.5 to 98.2]

ADVERSE EVENTS:
Time Frame: 15 minutes
Description: Regular monitoring by sponsor and mandatory reporting by investigator
Groups:
- Device Testing: As reported by user
Arm/Group | Device Testing
Serious Adverse Events (participants affected / at risk) | 0/206
Other Adverse Events (participants affected / at risk) | 0/206

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release.